CLINICAL TRIAL: NCT05368012
Title: MIDCAB (Mid-Calf Block) for Foot Surgery: A Pilot Study
Brief Title: MIDCAB (Mid-Calf Block) for Foot Surgery
Acronym: MIDCAB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-0066
Record Dates: First submitted 2022-03-29; First posted 2022-05-10 (Actual); Results first posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-02

CONDITIONS: Ankle Surgery; Foot Surgery
Keywords: foot and ankle surgery
MeSH Terms: interventions — Bupivacaine; Dexamethasone

STUDY DESIGN:
Intervention Model Description: All participants will receive the active MIDCAB block.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Active MIDCAB (Other): USG with a 25G needle, Bupivacaine 0.5% 30ml with 4mg preservative free dexamethasone divided as follows into the following 5 nerves: Posterior Tibial nerve (10ml), Saphenous nerve (5ml), Deep peroneal Nerve (5ml), Superficial peroneal nerve (5 ml), and Sural Nerve (5ml).
  Interventions: Drug: MIDCAB

INTERVENTIONS:
Drug: MIDCAB — Ultrasound-guided administration of the nerve block MIDCAB into mid-calf as analgesic intervention for patients.
  Other Names: Bupivacaine and dexamethasone

SUMMARY:
MIDCAB is defined as a group of ultrasound guided distal nerve blocks at the level of the individual branches. It is similar to an Ultrasound Guided (USG) Ankle block but the probe is placed higher on the calf covering all and any surgery of the foot and ankle, providing prolonged analgesia since we are blocking the individual nerves and preserving the proximal motor function.

This study is determining the potential therapeutic effect of MIDCAB during the hospital stay and recovery period in patients undergoing foot/ankle surgeries that require spinal anesthetic and peripheral nerve blocks. A total of 20 patients at HSS will participate to see if MIDCAB is not only effective at providing analgesia (pain relief) but to see if it allows allows patients to maintain motor function (movement) of the foot and ankle unlike the current popliteal block which is done above the knee and prevents patients from moving their foot.

During the course of the study we will also be looking at patients numeric pain scores with movement and at rest along with post-operative nausea and vomiting, the presence of numbness and it patients can move their foot. Along with all of these, the study will also look at the amount of opioid pain medications taken by patients along with medication-related side effects. As a result, the study will be used to determine if MIDCAB provides analgesia for patients undergoing foot/ankle surgery while allowing them to maintain movement of the foot. This pilot study will also be used to gather preliminary data that will allow us to perform a power analysis for a subsequent randomized clinical control trial that would compare the MIDCAB block to the popliteal block.

ELIGIBILITY:
Inclusion Criteria:

* Planned use of regional anesthesia
* Ability to follow the major components of the study protocol
* Planned foot or angle surgery

Exclusion Criteria:

* Patients younger than 18 years old and older than 80 years old
* Patients intending to receive general anesthesia
* Contra-indication to nerve blocks or spinal anesthesia
* Patients with an ASA status of IV or higher
* Chronic opioid use (taking opioids for longer than 3 months)
* Patients with prior foot or ankle surgery
* Patients with type 2 diabetes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Goytizolo, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article after de-identification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an Independent review committee ("learned intermediary") identified for this purpose and who have signed a DUA.

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: A total of 20 patients will be enrolled and will receive the stand of care analgesic protocol in addition to the following MIDCAB nerve block. There is only one treatment group in this study, no placebo group. The rationale behind there being one group is that this is a small pilot study that intends to inform subsequent randomized clinical control trials.
Period: Overall Study
Arm/Group | Treatment
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Active MIDCAB
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Block Duration
Description: The primary outcome will be block duration, how long the MIDCAB block provides analgesia. This will be measured via questionnaires of pain scores given to patients post surgical discharge (in PACU), 24h post surgical discharge, 48 hours post surgical discharge, and 1 week post surgical discharge. This will be done by measuring the change in patient's pains scores over the course of 7 days. Pain scores will be measured via NRS pain scale; the NRS (numeric rating scale) is a questionnaire that measures pain on a numeric scale, 0 (no pain) to 10 (worst pain imaginable). Patients will be asked to state the specific time-points they began to have pain after surgery.
Time Frame: Out to 1 week postoperatively
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Active MIDCAB
Number analyzed (Participants) | 20
hours | 18.2 [4.5 to 24.0]

2. Secondary Outcome: Number of Participants With Return of Motor Function of Foot and Ankle Post-Operatively
Description: The return of the patient's foot/ankle motor function which will be measured by whether the patient can dorsiflex/plantarflex at the ankle or have flexion/extension of the toes.
Time Frame: Measured in the PACU (post-anesthesia care unit) immediately upon patients arrival into the PACU, up to 1 hour after surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Active MIDCAB
Number analyzed (Participants) | 20
Participants | 20

3. Secondary Outcome: Cumulative Opioid Consumption
Description: Cumulative opioid consumption in morphine equivalents will be recorded post surgical discharge (in PACU), 24h post surgical discharge, 48 hours post surgical discharge, and 1 week post surgical discharge.
Time Frame: PACU (up until patients' discharge from the hospital), POD1 (Around 24 hrs after the PACU arrival time), POD2 (Around 48 hrs after the PACU arrival time) & POD7 (Around 1 week from the PACU arrival time)
Measure: Median (Inter-Quartile Range); unit: mg oral morphine equivalents
Arm/Group | Active MIDCAB
Number analyzed (Participants) | 20
mg oral morphine equivalents
  PACU | 0 [0 to 7.5]
  POD1 | 15 [0 to 33.8]
  POD2 | 8.8 [3.8 to 27]
  POD7 | 30 [7.5 to 67.5]

4. Secondary Outcome: Presence of Paresthesia (Numbness)
Description: Patients will be asked if they have any residual numbness in the foot or toes where the surgery took place.
Time Frame: POD 7 (1 week post-surgical discharge)
Measure: Count of Participants; unit: Participants
Arm/Group | Active MIDCAB
Number analyzed (Participants) | 20
Participants | 5

5. Secondary Outcome: Presence of Skin Irritation and Wounds
Description: Patients will be asked if they have any wounds or irritation to the skin (i.e. rashes, itching, burning, etc.) on the skin at the site of surgery and/or site of the block.
Time Frame: POD 7 (1 week post-surgical discharge)
Measure: Count of Participants; unit: Participants
Arm/Group | Active MIDCAB
Number analyzed (Participants) | 20
Participants | 2

6. Secondary Outcome: Presence of Nausea
Description: The questionnaire used asks patients if they have experienced any nausea.
Time Frame: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Active MIDCAB
Number analyzed (Participants) | 20
Participants
  PACU | 1
  POD1 | 2
  POD2 | 3
  POD7 | 2

7. Secondary Outcome: Severity of Nausea
Description: Patients are asked on a scale from 0-10 (0 being not severe and 10 being the worst severity) how severe their nausea was. This will be measured post surgical discharge (in PACU), 24h post surgical discharge, 48 hours post surgical discharge, and 1 week post surgical discharge
Time Frame: as for outcome 3
Population: The number analyzed is different than the overall number analyzed due to the fact that not every patient experienced any nausea. Only the patients who experienced nausea then got the follow up question about the severity of it.
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | Active MIDCAB
Number analyzed (Participants) | 20
Scores on a scale
  PACU: number analyzed (Participants) | 1
  PACU | 3 [3 to 3]
  POD1: number analyzed (Participants) | 2
  POD1 | 6.5 [6 to 7]
  POD2: number analyzed (Participants) | 3
  POD2 | 3.67 [2 to 5]
  POD7: number analyzed (Participants) | 2
  POD7 | 3 [3 to 3]

8. Secondary Outcome: Number of Total Episodes of Nausea
Description: Patients were asked how many episodes of nausea had occurred.
Time Frame: as for outcome 3
Population: as for outcome 7
Measure: Mean (Full Range); unit: episodes
Arm/Group | Active MIDCAB
Number analyzed (Participants) | 20
episodes
  PACU: number analyzed (Participants) | 1
  PACU | 1 [1 to 1]
  POD1: number analyzed (Participants) | 2
  POD1 | 2 [1 to 3]
  POD2: number analyzed (Participants) | 3
  POD2 | 1.33 [1 to 2]
  POD7: number analyzed (Participants) | 2
  POD7 | 1.5 [1 to 2]

ADVERSE EVENTS:
Time Frame: Adverse Event Data was collected for 7 days post surgery
Description: Adverse event collection was collected via phone call/patient reported
Arm/Group | Active MIDCAB
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-03): https://cdn.clinicaltrials.gov/large-docs/12/NCT05368012/Prot_SAP_000.pdf